CLINICAL TRIAL: NCT02869659
Title: Valued EpiGenetic Glycemic ImprovEments Through Weight Loss
Acronym: VEGGIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Medifast, Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00036970; R01DK103531 (NIH)
Record Dates: First submitted 2016-07-25; First posted 2016-08-17 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Obesity; Pre-diabetes
Keywords: obesity; pre-diabetes; overweight; lifestyle change; glucose
MeSH Terms: conditions — Obesity; Glucose Intolerance; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control/Delayed Weight Loss Group (Active Comparator): Control/Delayed Weight Loss Group: (18 weeks) Participants randomized to the delayed weight loss intervention (n=100) will serve as a no-weight loss control to the weight loss group during the first 18 weeks of the study. During the control (18 weeks) phase these participants will receive a monthly phone call visit from staff to maintain contact and interest in the study. At the end of the initial 18 weeks participants will complete all follow up assessments prior to being offered the opportunity to participate in a weight loss program.
  No outcome data will be collected at the end of the delayed weight loss phase.
  Interventions: Behavioral: Delayed Weight Loss
- Weight Loss Group (Experimental): Weight Loss group: Phase 1 (18 wks): Participants assigned to this group will undergo a dietary intervention for the first 18 weeks of the study.
  This level of weight loss will be achieved through the combination of a partial meal replacement (MR) program and individual and group nutrition/behavioral counseling. Participants will be provided with and asked to consume 4 Medifast® MR per day.
  Phase 2 (8 wks): After completion of the active weight loss phase, participants in this group will attend bimonthly group meetings to discuss increasing their activity.
  Phase 3 (26 wks): After completion of phase 2, participants will be called monthly for 26 weeks and then asked to return for a maintenance visit at the end of the 52 weeks from study start.
  Interventions: Behavioral: Weight Loss Group

INTERVENTIONS:
Behavioral: Weight Loss Group — All participants will follow the Medifast Achieve TM 4 & 2 & 1 Plan® which includes the 4 MR products per day, with the addition of 2 Lean and Green™ Meals and 1 Healthy Snack
  Arms: Weight Loss Group
Behavioral: Delayed Weight Loss — 18 weekly, group dietary and exercise sessions led by the study staff in which participants will follow a modified Diabetes Prevention Program
  Arms: Control/Delayed Weight Loss Group

SUMMARY:
This randomized controlled clinical trial will use methylomic and transcriptomic profiling to examine the effects of a weight loss intervention on the cholesterol metabolism gene network in monocytes and adipocytes and investigate the longitudinal relationship between these modifications and glycemic improvements.

DETAILED DESCRIPTION:
The investigators plan to recruit a total of 200 middle-aged (40-65 years) obese (BMI=30-39.9 kg/m2), sedentary, pre-diabetic participants who will be randomized to either a 18-week dietary weight loss (n=100) followed by a 8-week transition and then 26 weeks of maintenance (Weight Loss group) or a delayed weight loss (Control group, n=100) intervention.

During the screening visit, eligible participants who provided informed consent will complete a 3-day food record and then start a 3-day run-in period using the Medifast® meal replacement products to be used for the weight loss intervention. At the next visit the participant will meet with the Registered Dietitian (RD) to undergo an assessment of Readiness to Change (18). All participants must be approved for eligibility by the RD based on her clinical judgment of likelihood of success for weight loss, likelihood of compliance to the Medifast® meal plan, and willingness to be randomized to either group.

Control/Delayed Weight Loss Group: (18 weeks) Participants randomized to the delayed weight loss intervention (n=100) will serve as a no-weight loss control to the weight loss group during the first 18 weeks of the study. During the control (18 weeks) phase these participants will receive a monthly phone call visit from staff to maintain contact and interest in the study. At the end of the initial 18 weeks participants will complete all follow up assessments prior to being offered the opportunity to participate in a weight loss program. This weight loss program will involve 18 weekly, group dietary and exercise sessions led by the study staff in which participants will follow a modified Diabetes Prevention Program. Participants will be given an individual introduction session to the weight loss program by study staff and will be guided by the RD on their food purchasing and preparation of their meals, but no meal replacements or supplements will be provided.

Weight Loss group: Phase 1 (18 weeks): Participants assigned to this group will undergo a dietary intervention for the first 18 weeks of the study designed to elicit an approximate 8-10% weight loss. The intervention will incorporate partial meal replacements, nutrition education, and some behavior modification.

This level of weight loss will be achieved through the combination of a partial meal replacement (MR) program and individual and group nutrition/behavioral counseling. Participants will be provided with and asked to consume 4 Medifast® MR per day. All participants will follow the Medifast Achieve TM 4 & 2 & 1 Plan® which includes the 4 MR products per day, with the addition of 2 Lean and Green™ Meals and 1 Healthy Snack. The Lean and Green™ Meals will be prepared by the participants and each will consist of 5-7 oz. lean protein, 3 servings of non-starchy vegetables and up to 2 servings of healthy fat. The Healthy Snack will consist of one serving of fruit, dairy, or grain. Each MR from Medifast® contains ~90-110 kcals and 10-15 g protein. Participants will be given an individual introduction on the meal plan prior to starting and will be guided by the RD on their food purchasing and preparation of the other Lean and Green TM meals. They are encouraged to consume only what is approved on the Medifast Achieve TM 4 & 2 & 1 Plan®.

Phase 2 (8 weeks): After completion of the active weight loss phase, participants in this group will attend bimonthly group meetings to discuss increasing their activity. The goal is for participants to slowly increase their activity to 150 minutes per week and then continue at 150 minutes per week to help them maintain their weight. Activity logs will be dispensed and topics such as tracking activity, finding time for fitness and getting active will be discussed.

Participants will have the option to transition off the meal replacements and potentially continue on a select few during the transition phase. Additional dietary guidance will be available to help participants transition off MR and maintain their weight. The RD will calculate individual maintenance calorie goals to be discuss with participants at a brief individual session prior to starting the transition phase. At this session an introduction to the transition phase and information on how to track their activity will also be discussed.

Phase 3 (26 weeks): After completion of phase 2, participants will be called monthly for 26 weeks and then asked to return for a maintenance visit at the end of the 52 weeks from study start. Participants will be offered an optional session with a staff member at the time of their exit to discuss long term goals and strategies and provide closure.

ELIGIBILITY:
Inclusion Criteria:

* BMI=30-45.0 kg/m2 OR BMI 27-30, if waist circumference is ≥ 40in in men or ≥ 35in in women
* Sedentary for past 6 mos (<20 min; 2 d/wk of resistance or aerobic exercise)
* Normal cognitive function:

Greater than 12 years education:

Caucasian - MOCA ≥ 24 African American/Hispanic/Other- MOCA ≥ 22

12 years or less education: Caucasian- MOCA ≥22 African American/Hispanic/Other- MOCA ≥20

* No evidence of clinical depression
* Fasting blood glucose 100-125 mg/dl OR Hemoglobin A1c 5.7% - 6.4%
* No contraindications for participation in weight loss
* Able to provide own transportation to study visits and intervention
* Approved for participation by Medical Director
* Negative pregnancy test or confirmed post-menopausal/surgically sterile status (Women Only)
* Not involved in any other research study
* Willing to provide informed consent

Exclusion Criteria:

* Weight loss (±5%) in past 6 months
* Uncontrolled arrhythmias
* Cancer requiring treatment in past year, except non-melanoma skin cancers
* Regular smoker (>1 cigarette/day) or heavy drinker (>9 alcoholic drinks/wk) within past year
* Insulin dependent or uncontrolled diabetes (FBG>126 mg/dl) OR (Hemoglobin A1c 6.5% or greater)
* Uncontrolled hypertension (BP>160/90 mmHg)
* Elevated triglyceride (TG>400 mg/dl)
* Clinically evident liver disease, kidney disease, edema or anemia
* Past or current ischemic heart disease, uncontrolled angina, heart failure, PAD, stroke, chronic respiratory disease, endocrine or metabolic disease, neurological or hematological disease
* Regular use growth/steroid hormones, including estrogen replacement, weight loss medications, diabetes medications including insulin and/or blood thinners
* History of any type of bariatric or weight loss surgery or bilateral oophorectomy requiring long term hormone replacement therapy use

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Chang in Epigengene score (and related individual transcriptional and methylation measures) | baseline and 18 weeks
  The eigengene score is defined as the first principal component of a transcriptional network.

SECONDARY OUTCOMES:
change in glucose tolerance | baseline and 18 weeks
  A 2-hr OGTT will be performed to assess changes in glucose tolerance and insulin responses to the glucose challenge. Blood samples will be drawn before and after (30, 60, 90, and 120 min) a 75-g glucose ingestion for the determination of plasma glucose and insulin.
change in homeostatic model assessment (HOMA) estimates of insulin resistance | baseline and 18 weeks
  A 2-hr OGTT will be performed to assess changes in glucose tolerance and insulin responses to the glucose challenge. Blood samples will be drawn before and after (30, 60, 90, and 120 min) a 75-g glucose ingestion for the determination of plasma glucose and insulin. An estimate of insulin sensitivity by the homeostasis model assessment (HOMA) score will be calculated with the formula: fasting plasma insulin (μU/ml) × glucose (mmol/l)/22.5 (25). Glucose and insulin areas will be determined using Tai's model(26): ½×30×(y0min+2y30min+2y60min+2y90min+y120min), where y represents insulin or glucose values at the different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Jingzhong Ding, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mishra SP, Wang B, Jain S, Ding J, Rejeski J, Furdui CM, Kitzman DW, Taraphder S, Brechot C, Kumar A, Yadav H. A mechanism by which gut microbiota elevates permeability and inflammation in obese/diabetic mice and human gut. Gut. 2023 Oct;72(10):1848-1865. doi: 10.1136/gutjnl-2022-327365. Epub 2023 Mar 22. PMID 36948576

DOCUMENTS (1):
  • Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT02869659/ICF_000.pdf